CLINICAL TRIAL: NCT02264392
Title: Ultrasound Guided Versus Blind Incision and Drainage for the Treatment of Soft Tissue Abscesses in the Emergency Department
Brief Title: US Guided Versus BlindI&D for Treatment of Soft Tissue Abscesses in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Romolo Gaspari, Executive Vice Chair, Department of Emergency Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMASSEDUS4
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Abscess
MeSH Terms: conditions — Abscess | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Guided (Active Comparator): Ultrasound Guided Incision and Drainage- Patients will undergo ultrasound guided drainage of the abscess using bedside ultrasound
  Interventions: Procedure: Ultrasound Guided Incision and Drainage
- Blind I&D (Active Comparator): Blind Incision and Drainage- Patients will undergo drainage of the abscess using physical exam.
  Interventions: Procedure: Blind Incision and Drainage

INTERVENTIONS:
Procedure: Ultrasound Guided Incision and Drainage — Ultrasound guidance of the abscess drainage
  Arms: Ultrasound Guided
Procedure: Blind Incision and Drainage — Incision and drainage of abscess guided by physical exam alone
  Other Names: I&D
  Arms: Blind I&D

SUMMARY:
Standard treatment for a soft tissue abscess involves incision over the area of maximum fluctuance with drainage of purulence from the abscess cavity. The use of bedside ultrasound to guide this drainage has the potential to improve treatment outcomes by ensuring complete drainage of the cavity.

Our hypothesis is that the use of ultrasound for guidance of incision and drainage of soft tissue abscesses will decrease treatment failure rate compared to standard blind incision and drainage.

This hypothesis will be tested utilizing a blinded, randomized trial comparing standard incision and drainage to ultrasound guided incision and drainage.

DETAILED DESCRIPTION:
4) Background* The incidence of soft tissue infections is increasing, representing over 30 million emergency department visits per year. While there has been extensive research in recent years surrounding the use of antibiotics for soft tissue abscesses, the surgical management remains unchanged with standard therapy consisting of blind incision and drainage of the abscess cavity.

Despite incision and drainage and a spectrum of antibiotic coverage, treatment failure rates for these infections range from 5-20%. It is possible that part of this treatment failure can be attributed to inadequate abscess cavity evacuation. With blind drainage, it is possible that residual purulence or unforeseen satellite abscess cavities contribute to the persistence of the infection.

Ultrasound has been shown to aid in the identification of soft tissue abscesses and to help differentiate cellulitis from an abscess. Over the last decade, clinician performed bedside ultrasound has become a standard in the practice of emergency medicine with proficiency requirements now in place for graduating emergency medicine residents. While many practitioners have in fact adopted ultrasound in its use for the identification of abscesses, few subsequently use the ultrasound for procedural guidance.

We are specifically interested in studying the use of ultrasound for identifying the ideal location for initial incision as well as use of post procedural ultrasound to confirm complete evacuation of abscess purulence.

5) Inclusion and Exclusion Criteria*

Subjects enrolled in this study will include patients presenting to the emergency department with a diagnosis of soft tissue abscess. This includes patients of all ages and gender but will exclude individuals who cannot give consent or are prisoners (as they cannot return for follow up or be contacted for follow up).

Inclusion Criteria:

1. Soft tissue abscess suspected by patient history and physical exam and confirmed by bedside ultrasound
2. Able to provide written consent/ assent
3. Incision and drainage to be performed by ED physician

Exclusion Criteria:

1. Peritonsillar abscess
2. Pilonidal cyst, genital or perirectal abscess
3. Post-surgical wound infections
4. Pregnant
5. Prisoners
6. Previous incision and drainage for current abscess

6) Study-Wide Number of Subjects* N/A - Not a multi center study.

7) Study-Wide Recruitment Methods* Study subjects will be recruited from the patient population of the emergency departments on the Memorial and University campuses of UMASSMemorial Medical Center. Patients with signs and symptoms of soft tissue abscess confirmed by bedside ultrasound will be identified and enrolled by treating physicians. This will occur 24 hours a day, 7 days a week.

8) Study Timelines* A study subject's participation in the study will last for 1 week from the time of enrollment. This will consist of the initial study visit (emergency department encounter for treatment of the abscess), a follow-up visit at 2-3 days for wound evaluation and wick removal, and a telephone encounter at 1 week to 10 days.

Based on previous studies conducted by our group with a similar patient population and study protocol, we anticipate enrollment of 274 patients will take 2 years.

9) Study Endpoints*

The primary endpoint is failure of treatment at 7 days. This is defined as any of the following:

1. Need for repeat incision and drainage
2. Need for additional antibiotic coverage
3. Hospital Admission for intravenous antibiotics following the initial encounter 10) Procedures Involved* Patients presenting to the emergency department with suspected superficial abscesses that require an incision and drainage will be eligible for enrollment. Patients will be randomized into one of two groups: 1) Ultrasound Guided Incision and Drainage and 2) Standard Incision and Drainage. As a patient is identified for enrollment, the investigator will open a study packet containing standardized data collection sheet, consent documents and random designation for treatment group.

Group 1 Protocol: Ultrasound-guided Incision and Drainage Patients will be identified that require Incision and Drainage. An initial ultrasound will be performed to localize the abscess cavity. Anesthetic will be provided in the standard fashion by injected into the skin around the abscess. Incision of the skin overlying the abscess cavity and drainage of the purulent material will be followed by a repeat ultrasound to assess for complete drainage. Any additional pockets identified will be targeted for drainage until repeated ultrasound imaging demonstrates that the abscess cavity is completely drained. This post procedural ultrasound is performed on all patients currently undergoing ultrasound guided drainage of a superficial abscess. In patients where drainage cannot be completed, surgery will be consulted. The procedure will then be completed with placement of an iodoform wick and bulky dressing. Patients will be placed on oral antibiotics at the discretion of the treating attending physician and instructed to return in 2-3 days to the emergency department for re-evaluation and wick removal or sooner if problems arise. If necessary, additional drainage maybe performed. Additional I&D will be performed with or without ultrasound at the discretion of the attending physician.

A telephone follow-up 7-10 days post-procedure will be performed. Questions asked in follow up are located on the follow-up data sheet. See attachments or addendum. Blinding to the treatment group is accomplished by having follow up to determine the outcome of the treatment performed by an individual who is blinded to the initial ultrasound findings or treatment group.

Group 2 Protocol: Standard Incision and Drainage Patients will be identified that require Incision and Drainage*. Anesthetic will be provided in the standard fashion by injection in the skin around the abscess. Incision of the skin overlying the abscess cavity and drainage of the purulent material will be followed by placement of an iodoform wick and bulky dressing. Patients will be placed on oral antibiotics at the discretion of the treating attending physician and instructed to return in 2 days to the emergency department for re-evaluation and wick removal or sooner if problems arise. If necessary, additional drainage maybe performed. Additional I&D will be performed with or without ultrasound at the discretion of the attending physician.

A telephone follow-up 7 days post-procedure will be performed. This is the same follow up as in group 1. The research personnel will introduce themselves as research personnel from UMASS and will inform the subject that they are following up from their recent visit to the ED. They will ask the questions from the telephone follow-up data sheet and will refer to it as they conduct the follow up.

Blinding to the treatment group is accomplished by having follow up to determine the outcome of the treatment performed by an individual who is blinded to the initial ultrasound findings or treatment group.

*This decision may be made solely based on history and physical exam or by inital identification with ultrasound. If the presence of an abscess is initially identified without ultrasound, the original treating physician can continue to perform the Incision and Drainage procedure. If the presence of an abscess is initially identified with an ultrasound then another physician will need to perform the standard Incision and Drainage. The second physician is at liberty to perform the standard history and physical to assess the presence of the abscess prior to drainage. The second physician may be another resident or the attending physician overseeing the patient's care, provided they are blinded to the initial ultrasound identifying the presence of the abscess.

A standardized data sheet will record patient information, results of the procedure, time to perform the procedure, need for additional drainage and post-procedure recurrence of the abscess, need for change in oral antibiotic coverage and need for admission to the for intravenous antibiotics.

12) Data Management* Power Calcuation - Assuming an alpha of 0.05 and a beta of 0.2 and projected failure rate in the blind incision and drainage group of 20%, 119 subjects in each group will be required to detect a 20% reduction in treatment failure. Accounting for a 15% loss to follow-up will require a total number of subjects of 274 subjects. Patients assigned to each group will undergo analysis using the intention to treat principles.

Data will be stored on a password-protected computer in the locked offices of the department of emergency medicine on the University Campus of UMASSMemorial Medical Center. Only study personnel and the UMASS IRB will have access to the data.

Descriptive data will be analyzed using mean and standard deviation. Comparison between groups will be performed using Chi square analysis (categorical data) and Student's T-test (continuous data).

ELIGIBILITY:
Inclusion Criteria:

1. Soft tissue abscess suspected by patient history and physical exam and confirmed by bedside ultrasound
2. Able to provide written consent/ assent
3. Incision and drainage to be performed by ED physician

Exclusion Criteria:

1. Peritonsillar abscess
2. Pilonidal cyst, genital or perirectal abscess
3. Post-surgical wound infections
4. Pregnant
5. Prisoners
6. Previous incision and drainage for current abscess

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Failure of Therapy | 7 days
  Patient with a reoccurrence of the abscess

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD, PhD, Principal Investigator — UMass Memorial Health
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Gaspari RJ, Sanseverino A, Gleeson T. Abscess Incision and Drainage With or Without Ultrasonography: A Randomized Controlled Trial. Ann Emerg Med. 2019 Jan;73(1):1-7. doi: 10.1016/j.annemergmed.2018.05.014. Epub 2018 Aug 17. PMID 30126754